CLINICAL TRIAL: NCT00153413
Title: West Virginia WISEWOMAN Pilot Study to Test a Brief Nutrition Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDC-NCCDPHP-4114; U58/CCU322798-01 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Heart Disease; Blood Pressure; Obesity
MeSH Terms: conditions — Heart Diseases; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Masking Description: Participants are low income uninsured and underinsured so they must be masked.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Receive Cookin' Up Health, a nutrition intervention
  Interventions: Behavioral: Cookin' Up Health

INTERVENTIONS:
Behavioral: Cookin' Up Health — A brief nutrition intervention designed to improve dietary habits
  Other Names: Nutrition Intervention

SUMMARY:
To provide low-income, under- or uninsured 40- to 64-year-old women with the knowledge, skills, and opportunities to improve diet, physical activity, and other lifestyle behaviors to prevent, delay and control cardiovascular and other chronic diseases.

DETAILED DESCRIPTION:
To test whether a brief, interactive, computer-based nutrition intervention (Cookin' Up Health)impacts various health outcomes

ELIGIBILITY:
Inclusion Criteria:

* NBCCEDP
* Aged 40-64
* Attends selected rural clinics

Exclusion Criteria:

-

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Servings of fruits and vegetables | 3 months
  Based on food frequency questionnaire

SECONDARY OUTCOMES:
Ability to read food labels | 3 months
  Knowledge questions
Readiness to eat 5 fruits and vegetables per day | 3 months
  Based on Prochaska and DeClemente
Dietary Fat Score | 3 month
  Based on self-reported food frequency score

CONTACTS AND LOCATIONS:
Overall Officials: Julie Will, Study Chair — Centers for Disease Control and Prevention

REFERENCES:
- [Background] Santos L. The impact of nutrition and lifestyle modification on health. Eur J Intern Med. 2022 Mar;97:18-25. doi: 10.1016/j.ejim.2021.09.020. Epub 2021 Oct 17. PMID 34670680